CLINICAL TRIAL: NCT03399383
Title: Adherence and Perception With Hormone Replacement Therapy in Chronic Adrenal Insufficiency - Influence of a Standardized Patient Education
Brief Title: Adherence in Chronic Adrenal Insufficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: Medical University of Graz, Austria (Unknown); Medical practice for Endocrinology in Oldenburg, Germany (Unknown); Charite University, Berlin, Germany (Other); University Hospital, Frankfurt, Germany (Unknown); Endocrinology in Charlottenburg, Berlin, Germany (Unknown); University Hospital Munich, Germany (Unknown); University Hospital of Rostock, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Compliance-TRIAL
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Adrenal Insufficiency
Keywords: Adrenal Insufficiency; Adrenal crisis; Adherence; Standardized patient education
MeSH Terms: conditions — Adrenal Insufficiency | interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: Within the longitudinal part of the trial, patients with chronic adrenal insufficiency will be assessed by questionnaire before and after participation in the standardized education program (=intervention).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient education (longitudinal analysis) (Other): Patients with adrenal insufficiency complete a questionnaire before and 6 months after participation in a standardised patient education.
  Interventions: Other: Patient education

INTERVENTIONS:
Other: Patient education — Participation in the standardized education program (90min patient education). During sessions of 90-120 minutes duration, patients are educated in basic knowledge on adrenal insufficiency including the correct behaviour in emergency settings. Participants are provided with emergency cards and sets and are trained in self-injection of glucocorticoids.

SUMMARY:
Adherence, concerns and satisfaction with information in German patients with adrenal insufficiency as well as the influence of a standardized education program will be assessed by a compared cross-sectional and longitudinal study.

DETAILED DESCRIPTION:
Patients with adrenal insufficiency (AI) require a lifelong replacement therapy with glucocorticoids (GC). To avoid over- and under- replacement, an individual daily dose scheme and adequate dose adjustment during stressful events is essential. Recent patient surveys revealed nonadherence to treatment, concerns about GC and dissatisfaction with the provided information.

The aim of this trial is to evaluate the adherence, concerns and satisfaction with information in German patients with primary and secondary AI (PAI/SAI) and the influence of a standardized education program.

Patients with AI on GC therapy will be assessed by questionnaire, including the Medication Adherence Report Scale* (MARS), Beliefs about Medicines Questionnaire* (BMQ, adapted for AI) and Satisfaction with Information about Medicines Scale* (SIMS).*©Professor Rob Horne.

The study includes one cross-sectional-analysis and one longitudinal study (patient survey before and after participation at the standardized education program in Germany).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient's written informed consent
* Ability to comply with the protocol procedures
* Patients with chronic adrenal insufficiency under established stable replacement therapy

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Beliefs about Medicines Questionnaire (BMQ) | 6 months
  Evaluation of "Beliefs about Medicines" by BMQ-questionnaire (modified BMQ AI Specific© by Prof Rob Horne). The modified BMQ AI Specific© comprises: a 5-item Glucocorticoid-Necessity subscale assessing the participant's views about their personal need for the glucocorticoid medication and an 11-item Glucocorticoid-Concerns subscale assessing participants' concerns about the potential adverse consequences of taking glucocorticoids. For each BMQ statement, participants indicated their agreement on a 5-point Likert scale (range 1 = strongly disagree to 5 = strongly agree). GC-Necessity and GC-Concerns scores are computed by summing all subscale responses, then dividing by the number of items (range 1-5). Scores near five indicate high Necessity. Scores near one indicate high Concern.
Satisfaction with Information about Medicines Scale (SIMS) | 6 months
  Evaluation of "Satisfaction with Information about Medicines" by SIMS-questionnaire (Prof Rob Horne). Participants complete the SIMS© to indicate their satisfaction with the information they had received about their glucocorticoids. The SIMS has two subscales. The first assesses satisfaction with the information received about the Action and Usage of glucocorticoids (SIMS AU 9-items). The second assesses satisfaction with information about dealing with Potential Problems associated with glucocorticoids (SIMS PP 8-items). For each subscale item, participants state whether they were satisfied with the amount of information they had received (about right, none needed) or dissatisfied (too much, too little, none received). Subscale scores are calculated by counting the total number of 'satisfied' responses.
Medication Adherence Report Scale (MARS) | 6 months
  Evaluation of "Adherence" by MARS-questionnaire. Participants rate their adherence to glucocorticoids on an 8-item Medication Adherence Report Scale (MARS)© (Prof Rob Horne), modified for AI. Participants rate the frequency with which they perform each type of nonadherent behaviour on a 5-point scale (1=very to 5=never). Scores are summed to give a total score (range 8-40); higher scores indicate higher reported adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Wuerzburg, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hahner S, Spinnler C, Fassnacht M, Burger-Stritt S, Lang K, Milovanovic D, Beuschlein F, Willenberg HS, Quinkler M, Allolio B. High incidence of adrenal crisis in educated patients with chronic adrenal insufficiency: a prospective study. J Clin Endocrinol Metab. 2015 Feb;100(2):407-16. doi: 10.1210/jc.2014-3191. Epub 2014 Nov 24. PMID 25419882
- [Background] Hahner S, Loeffler M, Fassnacht M, Weismann D, Koschker AC, Quinkler M, Decker O, Arlt W, Allolio B. Impaired subjective health status in 256 patients with adrenal insufficiency on standard therapy based on cross-sectional analysis. J Clin Endocrinol Metab. 2007 Oct;92(10):3912-22. doi: 10.1210/jc.2007-0685. Epub 2007 Aug 7. PMID 17684047
- [Background] Lovas K, Loge JH, Husebye ES. Subjective health status in Norwegian patients with Addison's disease. Clin Endocrinol (Oxf). 2002 May;56(5):581-8. doi: 10.1046/j.1365-2265.2002.01466.x. PMID 12030907
- [Background] Chapman SC, Llahana S, Carroll P, Horne R. Glucocorticoid therapy for adrenal insufficiency: nonadherence, concerns and dissatisfaction with information. Clin Endocrinol (Oxf). 2016 May;84(5):664-71. doi: 10.1111/cen.12991. Epub 2016 Feb 15. PMID 26641418
- [Background] Tiemensma J, Andela CD, Pereira AM, Romijn JA, Biermasz NR, Kaptein AA. Patients with adrenal insufficiency hate their medication: concerns and stronger beliefs about the necessity of hydrocortisone intake are associated with more negative illness perceptions. J Clin Endocrinol Metab. 2014 Oct;99(10):3668-76. doi: 10.1210/jc.2014-1527. Epub 2014 Sep 16. PMID 25226291
- [Background] Horne R, Weinman J. Patients' beliefs about prescribed medicines and their role in adherence to treatment in chronic physical illness. J Psychosom Res. 1999 Dec;47(6):555-67. doi: 10.1016/s0022-3999(99)00057-4. PMID 10661603